CLINICAL TRIAL: NCT00005307
Title: Etiology of Blood Dyscrasias: Analysis of the International Agranulocytosis and Aplastic Anemia Study Data
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 3009; R01HL042524 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Anemia, Aplastic; Blood Disease; Agranulocytosis
MeSH Terms: conditions — Anemia, Aplastic; Hematologic Diseases; Agranulocytosis

SUMMARY:
To quantify the role of drugs and other factors in the etiology of agranulocytosis and aplastic anemia.

DETAILED DESCRIPTION:
BACKGROUND:

Agranulocytosis and aplastic anemia are rare but serious blood diseases that can be caused by drugs and other environmental factors. In 1980, there were only limited quantitative estimates of the risk between various exposures, particularly drugs, and the two dyscrasias. The data were collected in the IAAAS, a multicenter population-based case-control study conducted from 1980 to 1986 in eight regions. The study was funded by a pharmaceutical company to investigate a single hypothesis, but information was obtained on all drugs and on other factors, enabling a general investigation of the dyscrasias.

DESIGN NARRATIVE:

The study was for retrospective data analysis only. Standard case-control methods were used. In most instances, multivariate analysis was used to control confounding, especially by simultaneous use of other causal drugs. Adverse effects and the relative safety of drugs in relation to the two dyscrasias were documented. Because the IAAAS was population-based, incidence rates were provided directly, and excess risks were estimated for associated drugs. Such quantitative measures of association were generally unavailable. Among the drugs that were analyzed were various categories such as psychotropics, antihistamines, and cardiovascular drugs, and individual drugs such as allopurinol. Factors other than drugs were also evaluated, including exposure to radiation and chemicals such as benzene and insecticides, history of viral infection, and history of allergy and other conditions.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-04; Study Completion 1991-03 (Actual)

REFERENCES:
- [Background] Kelly JP, Kaufman DW, Shapiro S. Risks of agranulocytosis and aplastic anemia in relation to the use of cardiovascular drugs: The International Agranulocytosis and Aplastic Anemia Study. Clin Pharmacol Ther. 1991 Mar;49(3):330-41. doi: 10.1038/clpt.1991.37. PMID 1672513